CLINICAL TRIAL: NCT03185845
Title: The Appropriate Anticoagulation Duration for Chronic Obstructive Pulmonary Disease With Pulmonary Thromboembolism-- A National Multicenter, Prospective, Randomized, Controlled Clinical Trial
Brief Title: The Appropriate Anticoagulation Duration for Chronic Obstructive Pulmonary Disease With Pulmonary Thromboembolism
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Jianguo He, Chief of Pulmonary Vascular Disease Center, Chinese Academy of Medical Sciences, Fuwai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016YFC1304402B
Record Dates: First submitted 2017-06-12; First posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: COPD Exacerbation; PTE - Pulmonary Thromboembolism
MeSH Terms: conditions — Pulmonary Embolism | interventions — Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prolonged anticoagulation (Experimental): 3 months longer anticoagulation after regular treatment
  Interventions: Drug: Warfarin
- Regular anticoagulation (No Intervention): stop anticoagulation after regular treatment

INTERVENTIONS:
Drug: Warfarin — tailored dose according to international normalized ratio (INR) for 3 months
  Arms: Prolonged anticoagulation

SUMMARY:
Anticoagulation is the most important treatment for pulmonary thromboembolism (PTE). The thromboembolism risk is especially high in patients with chronic obstructive pulmonary disease (COPD) exacerbations. However, there's no agreement on the most appropriate duration of anticoagulation in COPD with PTE to balance the risk of recurrence of thrombosis and bleeding. This randomized, controlled trial aims to evaluate the risk and benefit of prolonged anticoagulation compared with the regular 3-month anticoagulation in COPD with PTE.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients due to chronic obstructive pulmonary disease exacerbation and diagnosed as newly developed pulmonary thromboembolism
* Regular anticoagulation for 3 months and got CT pulmonary angiography

Exclusion Criteria:

* Patients with major bleeding during prior anticoagulation
* Patients need long term anticoagulation to treat other diseases
* Patients unwilling to receive prolonged anticoagulation

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 392 (Estimated)
Dates: Start 2017-06-15 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Venous thromboembolism recurrence | 3 years
  recurrence rate in %

SECONDARY OUTCOMES:
Chronic obstructive pulmonary disease exacerbations | 3 year
  total times

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Chaoyang Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided